CLINICAL TRIAL: NCT03293173
Title: Biomarker Driven and Dose Intensified Chemoimmunotherapy With Early CNS Prophylaxis in Patients Less Than 65 Years With High Risk Diffuse Large B-Cell Lymphoma
Brief Title: Biomarker Driven Intensified ChemoImmunotherapy With Early CNS Prophylaxis
Acronym: Bio-CHIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Lymphoma Group (Network)
Collaborators: Helsinki University Central Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG-LBC-06
Record Dates: First submitted 2017-09-05; First posted 2017-09-26 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: DLBCL; Chemoimmunotherapy; High risk; CNS prophylaxis; Biomarker-driven
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: Stratification into group A (standard) or group B (experimental) based on biological risk factors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Biologically low risk group, R-CHOEP-14
  Interventions: Combination Product: R-CHOEP
- Group B (Experimental): Biologically high risk group, DA-EPOCH-R
  Interventions: Combination Product: DA-EPOCH-R

INTERVENTIONS:
Combination Product: R-CHOEP — rituximab, cyclophosphamide, doxorubicin, etoposide, vincristine, prednisone
  Arms: Group A
Combination Product: DA-EPOCH-R — dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, rituximab
  Arms: Group B

SUMMARY:
This study is testing whether stratification of the patients according to biological risk factors for different treatment groups will improve the outcome of patients with clinically high diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
For young clinically high-risk diffuse large B-cell lymphoma (DLBCL) patients the optimal therapy has not been established. Previous Nordic phase II studies, where dose-dense chemoimmunotherapy (R-CHOEP-14) with systemic CNS prophylaxis (HD-Mtx and HD-AraC) was given, demonstrated favorable outcome in comparison to historical controls. However, the patients with biological risk factors, such as translocation of bcl2 and myc oncogenes or and/or high BCL2 and MYC expression or deletion 17p and/or high P53 expression had significantly higher risk of death, as compared to patients without aberrations. The figures provide evidence for an unmet clinical need for the patients with biological risk factors, and underscore the importance of a clinical trial, where both biological and clinical risk factors play a role in the treatment planning.

In this trial treatment intensity varies according to presence or absence of biological risk factors. All patients receive a prephase medication consisting of prednisone and vincristine and two cycles of R-CHOP and high dose (HD) methotrexate. Subsequently, depending on the biological risk factors either four additional cycles of R-CHOEP (standard arm with no risk factors) or four dose adjusted R-EPOCH courses (experimental arm with risk factors) are given, followed by one course of high dose cytarabine (Ara-C) and R. R-CHOEP courses should be given with a two-week and R-EPOCH with a three-week interval.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 64 years
* Histologically confirmed CD20+ DLBCL based on revised WHO 2008 Lymphoma Classification. The following subgroups and variants can be included:

  * ALK-positive large B-cell lymphoma
  * Intravascular large B-cell lymphoma
  * T-cell rich B-cell lymphoma
  * Myc/BCL-2 double hit lymphoma
  * Follicular lymphomas grade 3b
  * DLBCL with previously undiagnosed concurrent small cell infiltration in bone marrow, lymph node, or extranodal site and lymphomas intermediate between DLBCL and Burkitt's lymphoma are allowed
  * Posttransplantation lymphoma (PTLD), discordant or transformed lymphoma are NOT allowed
* Patients in at least stage II with age adjusted IPI score of 2 or 3:

  * Stage III /IV and elevated LDH
  * Stage III/IV and WHO performance status 2 - 3
  * Stage II and elevated LDH and WHO performance status 2 - 3
* And/or patients with site specific risk factors for CNS recurrence defined as follows

  * More than one extranodal site
  * Testicular lymphoma, stage IIE and higher
  * Paranasal sinus and orbital lymphoma with destruction of bone
  * Large cell lymphoma infiltration of the bone marrow
* Previously untreated, except steroids allowed
* WHO performance status 0-3
* Written informed consent

Exclusion Criteria:

* Severe cardiac disease: cardiac function grade 3-4, left ventricular ejection fraction <45%
* Impaired bone marrow liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule (Hemoglobin < 9 g/dL, ANC < 1.5 × 109/L, Platelet count < 75 × 109/L, creatinine clearance < 40 mL/min, ALT/AST > 2.5 x ULN, bilirubin 1.5 x ULN, INR > 1.5)
* Pregnancy/lactation
* Men and women of reproductive potential not agreeing to use effective contraception during treatment and for 18 months after completion of treatment (Effective contraception is combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), hormone-releasing IUD, bilateral tubal occlusion, vasectomised partner, or sexual abstinence
* Patients with other severe medical problems, including active infections, cardiac or pulmonary disease, history of PML and with an expected short survival for non-lymphoma reasons
* Known HIV positivity
* Active or chronic hepatitis B virus (HBV) infection (defined as positive HBsAg serology), or active hepatitis C virus (HCV) infection (defined by antibody serology testing). HBsAg, HBcAb, and HCVAb must be tested during screening. Patients who have protective titers of HBsAb along negative HBsAg after vaccination or prior but cured hepatitis B are eligible.
* Vaccination with a live vaccine within one month prior to randomization
* Patients with a malignancy that has been treated but not with curative intent, unless the malignancy has been in remission without treatment for ≥ 5 years prior to enrollment
* Earlier treatment containing anthracyclines
* Psychiatric or mental disorder which make the patient unable to give an informed consent and/or adhere to the protocol
* CNS disease as diagnosed by MRI or CSF cytology. Positive CSF flow cytometry below diagnostic threshold level by cytology is allowed
* Transformed lymphoma
* Primary mediastinal B-cell lymphoma
* Pleural or peritoneal fluid that cannot be drained safely
* Hypersensitivity to the active substance or any of the other ingredients
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Patients participating in other clinical studies, unless followed for survival
* Lower urinary tract constriction, which cannot be treated adequately
* Degenerative and toxic encephalopathy
* Neuromuscular disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) of the patients with biological risk factors | At 3 years
  Interval between the registration date and the date of documented progression or lack of response, first relapse, death for any reason or discontinuation/change of therapy because of toxicity, whichever occurs first. Otherwise, patients will be censored at the last date they were known to be alive. For patients not responding at any time point on study treatment, TTF is defined as one day.

SECONDARY OUTCOMES:
Time to treatment failure (TTF) at 3 years from date of registration of all patients and the patients in the low risk group | At 3 years
  Interval between the registration date and the date of documented progression or lack of response, first relapse, death for any reason or discontinuation/change of therapy because of toxicity, whichever occurs first. Otherwise, patients will be censored at the last date they were known to be alive. For patients not responding at any time point on study treatment, TTF is defined as one day.
Incidence of treatment-emergent adverse events (Safety and tolerability) | During the treatment period at the end of each cycle (14 or 21 days) up to 6 months. In addition, severe late toxicities during follow-up at 6 months intervals through study completion, an average of 5.5 years.
  Number of patients with treatment-related adverse events graded according to the NCI CTCAE v 4.03
Clinical response rate of all patients and the patients with biological risk factors | At the end of treatment cycles 2 and 7. Each cycle is two (group A) or three weeks (group B)
  Number of patients with complete or partial response
CNS relapse rate | At 1,5 years
  Number of patients with CNS progression
Progression free survival rate (PFS) of all patients and the patients with biological risk factors | At 3 years
Overall survival rate (OS) of all patients and the patients with biological risk factors | At 3 years
Molecular correlates for survival | At 3 years
  Identification of genomic aberrations (for example mutations and translocations), gene expression profiles and protein expression from the tumor tissue and circulation that predict clinical course of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Sirpa Leppa, prof, Principal Investigator — Helsinki University Hospital Cancer Centre
Locations (16):
- Denmark (5):
  - Aarhus University Hospital, Aarhus
  - Dept of Haematology, Rigshospitalet, Copenhagen
  - Dept of Haematology, Herlev Hospital, Copenhagen, Herlev
  - Dept haematology, Odense University hospital, Odense
  - Dept of Haematology, Sjaellands University hospital, Roskilde, Roskilde
- Finland (5):
  - Helsinki University Hospital Cancer Centre, Helsinki
  - Keski-Suomen keskussairaala, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - TAYS, Tampere
  - Turku University Hospital, Syöpäklinikka, Turku
- Norway (5):
  - Dept. of Oncology, Helse Bergen HF Haukeland sykehus, Bergen
  - Oslo University Hospital, Oslo
  - Dept. of Haematology and Oncology, Helse Stavander HF sykehuset, Stavanger
  - Dept. of Oncology, Universitetssykehuset i Nord-Norge HF, Tromsø
  - Dept of Oncology, St. Olavs hospital HF, Trondheim
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
individual deidentified participant data (including data dictionaries) will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Fiskvik I, Beiske K, Delabie J, Yri O, Spetalen S, Karjalainen-Lindsberg ML, Leppa S, Liestol K, Smeland EB, Holte H. Combining MYC, BCL2 and TP53 gene and protein expression alterations improves risk stratification in diffuse large B-cell lymphoma. Leuk Lymphoma. 2015 Jun;56(6):1742-9. doi: 10.3109/10428194.2014.970550. Epub 2014 Nov 19. PMID 25284491
- [Background] Holte H, Leppa S, Bjorkholm M, Fluge O, Jyrkkio S, Delabie J, Sundstrom C, Karjalainen-Lindsberg ML, Erlanson M, Kolstad A, Fossa A, Ostenstad B, Lofvenberg E, Nordstrom M, Janes R, Pedersen LM, Anderson H, Jerkeman M, Eriksson M. Dose-densified chemoimmunotherapy followed by systemic central nervous system prophylaxis for younger high-risk diffuse large B-cell/follicular grade 3 lymphoma patients: results of a phase II Nordic Lymphoma Group study. Ann Oncol. 2013 May;24(5):1385-92. doi: 10.1093/annonc/mds621. Epub 2012 Dec 17. PMID 23247661
- [Derived] Arffman M, Meriranta L, Autio M, Holte H, Jorgensen J, Brown P, Jyrkkio S, Jerkeman M, Drott K, Fluge O, Bjorkholm M, Karjalainen-Lindsberg ML, Beiske K, Pedersen MO, Leivonen SK, Leppa S. Inflammatory and subtype-dependent serum protein signatures predict survival beyond the ctDNA in aggressive B cell lymphomas. Med. 2024 Jun 14;5(6):583-602.e5. doi: 10.1016/j.medj.2024.03.007. Epub 2024 Apr 4. PMID 38579729